CLINICAL TRIAL: NCT00225160
Title: A Randomised Double Blinded Placebo Controlled Pilot Study to Evaluate the Safety and Efficacy of Acetyl L Carnitine in Combination With Antiretroviral Therapy for the Prevention of Distal Symmetric Polyneuropathy and Lipid Abnormalities in Treatment naïve HIV Infected Subjects
Brief Title: ALCAR Prophylaxis Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Free Hampstead NHS Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sigma-Tau Research, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALCAR
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections; Distal Symmetric Polyneuropathy
Keywords: HIV; poly neuropathy; acetyl L-carnitine; treatment naïve; combination antiretroviral therapy; Lipid abnormalities
MeSH Terms: conditions — HIV Infections | interventions — Acetylcarnitine

INTERVENTIONS:
Drug: acetyl L-carnitine

SUMMARY:
The purpose of this study is to determine whether Acetyl L-carnitine can prevent the development of nerve damage, known as neuropathy, in individuals taking anti-HIV drugs over a 48-week period. In addition the safety and tolerability of Acetyl L-carnitine will be assessed.

This study compares the use of Acetyl L-carnitine or placebo (a dummy drug) in the prevention of nerve damage. The current standard of care is to use painkillers to manage the pain, with little or no effect. The possible beneficial effects of taking Acetyl L-carnitine is to prevent nerve damage as a result of anti-HIV medication.

The main purposes of the trial are:

* to look at the differences in between those on Acetyl L-carnitine versus those on placebo
* to look at the effect on state of your nervous system in the two treatment groups by measuring nerve activity
* to learn more about the safety and tolerance of Acetyl L-carnitine

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged > 18 years of age
* HIV-1 infected as documented by a licensed HIV-1 antibody ELISA
* Women of childbearing potential must have a negative serum (beta-HCG; performed by a medical doctor - Austria only) pregnancy test within 28 days of starting study drug (and at monthly intervals for the duration for the trial (-Austria only)
* Ability to assess level of pain and complete a pain log
* Ability to understand and provide written informed consent to participation in this trial
* All clinical laboratory values must be considered not clinically significant - for the potential response to the planned new regimen - in the opinion of the investigator
* Naïve to antiretroviral therapy

Exclusion Criteria:

* Diminished ankle reflexes (compared to the knee) or absent ankle reflexes. OR
* Distal diminution of either vibration sense in the legs (defined as perception vibration < 10 seconds at the great toe with a tuning fork initially struck hard enough to be audible) or pain or temperature sensation.
* Subjects who in the investigator's opinion are unlikely to complete the 48 weeks trial period.
* Subjects with current alcohol or illicit drug use which, in the opinion of the investigator, may interfere with the subjects' ability to comply with the dosing schedule and protocol evaluations.
* Previous treatment with any drug known to induce peripheral neuropathy, specifically excessive alcohol, isoniazid & vincristine.
* Subjects with insulin dependent diabetes or cancer and an existing peripheral neuropathy or hereditary neuropathy.
* Subjects with Vitamin B 12 deficiency (level < 150pg/mL)
* Subjects using neurotoxic systemic therapeutic agents, systemic corticosteroids or immunomodulators within 30 days of randomisation.
* Use of a medication for neuropathic pain during 2 weeks prior to randomisation (including tricyclic antidepressants, mexilitene, phenytoin or carbamazepine).
* Subjects who have taken L-carnitine within 6 last months, or who have ever taken ALCAR.
* Subjects being pregnant or breast feeding.
* Subjects suffering from a serious medical condition, including one or more AIDS defining events (Appendix 8), which in the opinion of the investigator, would compromise the safety of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-11

PRIMARY OUTCOMES:
The change from baseline in total area of Protein Gene Product (PGP) immunostaining on the epidermis at 48 weeks

SECONDARY OUTCOMES:
-Proportion of patients requiring analgesic agents
-Changes in the global assessments of pain by both subject and investigator
-Proportion of patients with HIV-1 RNA < 50 copies/ml at 24 and 48 weeks
-Proportion of patients with virological failure at 24 and 48 weeks
-Changes in CD4+ cell count from baseline after 24 and 48 weeks of treatment
-Time to discontinuation of the randomised treatment and reasons for this
-Incidence of adverse events
-Incidence of clinical disease progression
-Proportion of patients at Weeks 24 and 48 and incidence of virological and clinical failure or treatment-limiting adverse events
-Proportion of patients with changes in lipid profiles
-Change in body habitus as measured by lipodystrophy questionnaire
-Change in QOL at Weeks 24 and 48
-Changes in subcutaneous adipose tissue mtDNA

CONTACTS AND LOCATIONS:
Overall Officials: Armin - Rieger, MD, Principal Investigator — University of Vienna Medical School AKH
Locations (1):
- Royal Free Hospital, London, United Kingdom